CLINICAL TRIAL: NCT03967756
Title: Impact of Automatic Polyp Detection System on Adenoma Detection Rate-a Multicenter,Prospective, Randomized Controlled Trial
Brief Title: Impact of Automatic Polyp Detection System on Adenoma Detection Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); Wenzhou Central Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-2
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Colonic Polyps; Colorectal Adenomas
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted withdrawal group (Experimental): A deep learning-based automatic polyp detection system was used to assist the endoscopist.
  Interventions: Device: Automatic polyp detection system
- Routine withdrawal group (No Intervention): Routine withdrawal without any assist.

INTERVENTIONS:
Device: Automatic polyp detection system — When colonoscopists withdraw the colonoscopies and inspect the colons, the video streaming of colonoscopies was real-time switched to the automatic polyp detection system, which made it feasible to detect lesions in real time. When any potential polyp is detected by the system， there will be a tracing box on an adjacent monitor to locate the lesion with a simultaneous sound alarm.
  Arms: AI-assisted withdrawal group

SUMMARY:
In recent years, with the continuous development of artificial intelligence, automatic polyp detection systems have shown its potential in increasing the colorectal lesions. Yet, whether this system can increase polyp and adenoma detection rates in the real clinical setting is still need to be proved. The primary objective of this study is to examine whether a combination of colonoscopy and a deep learning-based automatic polyp detection system is a feasible way to increase adenoma detection rate compared to standard colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40-85 years old who have indications for screening, surveillance and diagnostic.
* Patients who have signed inform consent form.

Exclusion Criteria:

* Patients who have undergone colonic resection
* Patients with intracranial and/or central nervous system disease, including cerebral infarction and cerebral hemorrhage.
* Patients with severe chronic cardiopulmonary and renal disease.
* Patients who are unwilling or unable to consent.
* Patients who are not suitable for colonoscopy
* Patients who received urgent or therapeutic colonoscopy
* Patients with pregnancy, inflammatory bowel disease, polyposis of colon, colorectal cancer, or intestinal obstruction
* Patients who are taking aspirin, clopidogrel or other anticoagulants
* Patients with withdrawal time < 6 min

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1118 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate(ADR) | 30 minutes
  the number of patients with at least one adenoma divided by the total number of patients.

SECONDARY OUTCOMES:
polyp detection rate(PDR) | 30 minutes
  the number of patients with at least one polyp divided by the total number of patients.
adenoma per colonoscopy | 30 minutes
  the number of adenomas detected during colonoscopy withdraw divided by the number of colonoscopies.
polyp per colonoscopy | 30 minutes
  the number of polyps detected during colonoscopy withdraw divided by the number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urban G, Tripathi P, Alkayali T, Mittal M, Jalali F, Karnes W, Baldi P. Deep Learning Localizes and Identifies Polyps in Real Time With 96% Accuracy in Screening Colonoscopy. Gastroenterology. 2018 Oct;155(4):1069-1078.e8. doi: 10.1053/j.gastro.2018.06.037. Epub 2018 Jun 18. PMID 29928897
- [Background] Ahmad OF, Soares AS, Mazomenos E, Brandao P, Vega R, Seward E, Stoyanov D, Chand M, Lovat LB. Artificial intelligence and computer-aided diagnosis in colonoscopy: current evidence and future directions. Lancet Gastroenterol Hepatol. 2019 Jan;4(1):71-80. doi: 10.1016/S2468-1253(18)30282-6. Epub 2018 Dec 6. PMID 30527583